CLINICAL TRIAL: NCT03262896
Title: Neurophysiological Study in Patients With Brain Death: A Single Center Prospective Study
Brief Title: Neurophysiological Examination in Patients With Brain Death
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Hilmi Demirkiran, MD, Assistant Professor, Yuzuncu Yil University
Other Study IDs: EMG in Brain Death
Record Dates: First submitted 2017-08-19; First posted 2017-08-25 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Brain Death
Keywords: Brain Death; Spinal Reflex; Electromyography
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with brain death: Ten patients with definite etiology, who were diagnosed with brain death because of Apnea test positive and / or cranial reflexes were not available and were male and female patients aged 18-72 years

SUMMARY:
This study examines muscle movements of elecromyography in adults with brain death. Half of the participants will have brain death, the other half will be healthy volunteers.

DETAILED DESCRIPTION:
In some of the patients who have brain death diagnosis, some movements may be seen. Because of these movements, the doctors sometimes avoid to make brain death diagnosis. So making brain death diagnosis may delay. And in these patients, even if the brain death diagnosis made the family members refuse to donate the organs of the patients because they think their patients may survive when they see muscle movements with touch. These patients with brain death are lost in a short time, so some of the patients can not be used as donors. In this study, the investigators aim to raise awareness the movements in brain death patients can be seen, to study the movements neurophysiologically by EMG, whether EMG can be used as auxiliary method or not in brain death diagnosis and to raise organ donation numbers from cadavers. Investigators will examine the motor response and F response in the facial nerve, median nerve, and tibialis posterior nerve with electromyography neurophysiologically.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with definite diagnosis of brain death,
* Patients with permission from their parents,
* Patients without trauma of medullaspinalis and peripheral nerve injuries,
* Patients without previously known muscle disease (Myasthenia gravis, myopathy, etc.),
* Patients with previously unknown neurological disease (Amyotrophic Lateral Sclerosis, Multiple sclerosis, Guillain Barre syndrome, Poliomyelitis, etc.),
* Patients who have not previous systemic diseases (Connective Tissue Disease, Diabetes mellitus, Chronic renal failure, etc.).

Exclusion Criteria:

* Uncertain brain death,
* Patients without permission of family members,
* Younger than 18 years old and older than 72 years,
* Patients with medulla spinalis and peripheral nerve injuries,
* Patients with known muscle disease (Myasthenia gravis, myopathy, etc.),
* Patients with neurological disease (Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Guillain Barre Syndrome, Poliomyelitis, etc.),
* Patients with previous systemic diseases (Connective Tissue Disease, Diabetes, Chronic Kidney Failure, etc.)

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the adult intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Axonal response | Within 72 hours from brain death diagnosis
  Measure of axonal response by electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Hilmi Demirkiran, MD, Study Director — Department of Anethesiology and Reanimation; Aydin Cagac, MD, Principal Investigator — Department of Neurology
Locations (1):
- Yuzuncu Yil University, School of Medicine, Van, Tusba / Zeve Kampus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided